CLINICAL TRIAL: NCT05431478
Title: Clinical Performance of Two Reusable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLL949-E005
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-09

CONDITIONS: Refractive Errors
Keywords: Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID022821, then AOHP (Other): Serafilcon A contact lenses worn during Period 1, with senofilcon A contact lenses worn during Period 2, as randomized. Each study lens type will be worn bilaterally (in both eyes) at least 10 hours per day for approximately 14 days. CLEAR CARE will be used for daily cleaning and disinfection. The serafilcon A contact lenses will be replaced with a fresh pair at the Week 1 follow-up visit.
  Interventions: Device: Serafilcon A contact lenses; Device: Senofilcon A contact lenses; Device: CLEAR CARE
- AOHP, then LID022821 (Other): Senofilcon A contact lenses worn during Period 1, with serafilcon A contact lenses worn during Period 2, as randomized. Each study lens type will be worn bilaterally (in both eyes) at least 10 hours per day for approximately 14 days. CLEAR CARE will be used for daily cleaning and disinfection. The serafilcon A contact lenses will be replaced with a fresh pair at the Week 1 follow-up visit.
  Interventions: Device: Serafilcon A contact lenses; Device: Senofilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Serafilcon A contact lenses — Reusable silicone hydrogel contact lenses worn during the day and removed at night for daily cleaning and disinfection
  Other Names: LID022821
Device: Senofilcon A contact lenses — Reusable silicone hydrogel contact lenses worn during the day and removed at night for daily cleaning and disinfection
  Other Names: ACUVUE OASYS® 2 Week with HYDRACLEAR® PLUS; AOHP
Device: CLEAR CARE — Hydrogen peroxide based contact lens cleaning and disinfecting solution
  Other Names: CLEAR CARE® Cleaning and Disinfecting Solution

SUMMARY:
The purpose of this study is to assess the clinical performance of two reusable silicone hydrogel contact lenses when worn on a daily wear basis.

DETAILED DESCRIPTION:
In this crossover study, subjects will wear each study lens type for approximately 14 days and attend 7 scheduled visits. The expected duration of subject participation in the study is approximately 28 days (approximately 14 days per each study lens type).

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.
* Best Corrected Visual Acuity of 20/25 Snellen (0.10 logMAR) or better in each eye.
* Willing to stop wearing habitual contact lenses for the duration of study participation.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any eye infection, inflammation, abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator.
* Habitual wear of AOHP contact lenses.
* Habitual wear of any daily disposable contact lenses.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Drs. Giedd, PA, Maitland, Florida
  - Wesley Optometric Consulting, Medina, Minnesota
  - ProCare Vision Center, Granville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all enrolled participants/eyes (68/136).
Units Other Than Participants: eyes
Groups:
- LID022821, Then AOHP: Serafilcon A contact lenses worn during Period 1, with senofilcon A contact lenses worn during Period 2, as randomized. Each study lens type was worn bilaterally (in both eyes) at least 10 hours per day for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection. The serafilcon A contact lenses were replaced with a fresh pair at the Week 1 follow-up visit.
- AOHP, Then LID022821: Senofilcon A contact lenses worn during Period 1, with serafilcon A contact lenses worn during Period 2. Each study lens type was worn bilaterally (in both eyes) at least 10 hours per day for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection. The serafilcon A contact lenses were replaced with a fresh pair at the Week 1 follow-up visit.
Period: Period 1, Approximately 14 Days
Arm/Group | LID022821, Then AOHP | AOHP, Then LID022821
Started | 34; 68 eyes | 34; 68 eyes
Completed | 34; 68 eyes | 34; 68 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Period 2, Approximately 14 Days
Arm/Group | LID022821, Then AOHP | AOHP, Then LID022821
Started | 34; 68 eyes | 34; 68 eyes
Completed | 34; 68 eyes | 34; 68 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- AOHP, Then LID022821: Senofilcon A contact lenses worn during Period 1, with serafilcon A contact lenses worn during Period 2, as randomized. Each study lens type was worn bilaterally (in both eyes) at least 10 hours per day for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection. The serafilcon A contact lenses were replaced with a fresh pair at the Week 1 follow-up visit.
- Total: Total of all reporting groups
Arm/Group | LID022821, Then AOHP | AOHP, Then LID022821 | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (7.1) | 30.9 (6.5) | 32.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 32 | 33 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 34 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity With Study Lenses at Week 1 Follow-Up
Description: Visual acuity (VA) was assessed with study lenses in place using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity. Each eye was assessed individually. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Week 1, each wear period. A wear period was approximately 14 days.
Population: Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID022821: Serafilcon A contact lenses worn during Period 1 or Period 2, as randomized, in both eyes at least 10 hours per day for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection. The serafilcon A contact lenses were replaced with a fresh pair at the Week 1 follow-up visit.
- AOHP: Senofilcon A contact lenses worn during Period 1 or Period 2, as randomized, in both eyes at least 10 hours per day for approximately 14 days. CLEAR CARE was used for daily cleaning and disinfection.
Arm/Group | LID022821 | AOHP
Number analyzed (Participants) | 68 | 68
Number analyzed (eyes) | 136 | 136
logMAR | -0.12 (0.07) | -0.11 (0.08)

ADVERSE EVENTS:
Time Frame: Adverse Events (AE's) were collected from time of consent to study exit, approximately 28 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AE's is reported in units of eyes; all other populations are reported in units of subjects.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID022821 Ocular; LID022821 Non-Ocular: Events reported in this group occurred while exposed to the serafilcon A contact lenses
- AOHP Ocular; AOHP Non-Ocular: Events reported in this group occurred while exposed to the senofilcon A contact lenses
Arm/Group | Pretreatment | LID022821 Ocular | LID022821 Non-Ocular | AOHP Ocular | AOHP Non-Ocular
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/136 | 0/68 | 0/136 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/136 | 0/68 | 0/136 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/136 | 0/68 | 0/136 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05431478/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT05431478/SAP_001.pdf